CLINICAL TRIAL: NCT01216683
Title: A 3-Arm Randomized Phase II Trial of Bendamustine-Rituximab (BR) Followed by Rituximab vs Bortezomib-BR (BVR) Followed by Rituximab vs BR Followed by Lenalidomide/Rituximab in High Risk Follicular Lymphoma
Brief Title: Bendamustine Hydrochloride and Rituximab With or Without Bortezomib Followed by Rituximab With or Without Lenalidomide in Treating Patients With High-Risk Stage II, Stage III, or Stage IV Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2408; E2408 (Other: ECOG-ACRIN); NCI-2011-02644 (Other: NCI); CDR0000683312 (Other: NCI)
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Rituximab; Bendamustine Hydrochloride; Bortezomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A then Arm D (Induction with Bendamustine + Rituximab; Continuation with Rituximab) (Experimental): Arm A (induction): Patients receive rituximab intravenously (IV) on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Arm D (continuation): Beginning 4 weeks after the completion of induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: Bendamustin
- Arm B then Arm E (Induction with Bendamustine + Rituximab + Bortezomib; Continuation with Rituximab) (Experimental): Arm B (induction): Patients receive rituximab IV on day 1; bortezomib IV on days 1, 4, 8, and 11; and bendamustine hydrochloride IV over 1 hour on days 1 and 4. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Arm E (continuation): Beginning 4 weeks after the completion of induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab as in arm D.
  Interventions: Biological: rituximab; Drug: Bendamustin; Drug: bortezomib
- Arm C then Arm F (Induction with Bendamustine+Rituximab; Continuation with Lenalidomide + Rituximab) (Experimental): Arm C (induction): Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Arm F (continuation): Immediately after completing induction therapy, patients who have stable disease or better at time of post-induction restaging receive oral lenalidomide on days 1-21. Treatment repeats every 4 weeks for 13 courses in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after the completion of induction therapy, these patients receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: Bendamustin; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; Chimeric anti-CD20 monoclonal antibody; Rituxan
Drug: Bendamustin — Given IV
  Other Names: Bendamustine hydrochloride; CEP-18083; TREANDA
Drug: bortezomib — Given IV
  Other Names: MLN341; LDP-341; Velcade®; PS-341
  Arms: Arm B then Arm E (Induction with Bendamustine + Rituximab + Bortezomib; Continuation with Rituximab)
Drug: lenalidomide — Given orally
  Other Names: IMiD compound CC-5013; Revlimid®
  Arms: Arm C then Arm F (Induction with Bendamustine+Rituximab; Continuation with Lenalidomide + Rituximab)

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. It is not yet known whether giving bendamustine hydrochloride and rituximab together alone is more effective than giving bendamustine hydrochloride and rituximab together with bortezomib or lenalidomide in treating follicular lymphoma.

PURPOSE: This randomized phase II trial is studying giving bendamustine hydrochloride and rituximab together with or without bortezomib followed by rituximab with or without lenalidomide to see how well they work in treating patients with high-risk stage II, stage III, or stage IV follicular lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the complete remission rate in patients with high-risk follicular lymphoma receiving induction therapy comprising bendamustine hydrochloride and rituximab with vs without bortezomib.
* To compare the 1-year post-induction disease-free survival rate in patients receiving continuation therapy comprising rituximab with vs without lenalidomide.

Secondary

* To determine the 3-year progression-free survival and the 5-year overall survival of these patients.
* To evaluate patient-reported outcomes at baseline and during treatment to determine differences in symptom palliation, treatment-related symptoms, and overall health-related quality of life.
* To examine the association between baseline Follicular Lymphoma International Prognostic Index (FLIPI) information and outcome of these patients.
* To examine the association between baseline and end-of-treatment patient comorbidities assessed by the Cumulative Illness Rating Scale (CIRS) and outcome.
* To create an image and tissue bank including serial PET/CT scans, diagnostic paraffin-embedded tissue, germline DNA, and serial blood and bone marrow samples sufficient to support proposed and future studies of tumor and host characteristics that may predict for clinical outcome, including treatment arm effects, and enhance existing prognostic indices. (exploratory)
* To evaluate the rate of peripheral neuropathy associated with subcutaneous and intravenous bortezomib.

OUTLINE: Patients are stratified according to FLIPI-1score (0-2 vs 3 vs 4-5) and Groupe d'Etude des Lymphomes Folliculaires (GELF) tumor burden (low vs high). Patients are randomized to 1 of 3 treatment arms.

* Arm A then Arm D

  * Arm A (induction): Patients receive rituximab intravenously (IV) on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Arm D (continuation): Beginning 4 weeks after the completion of induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
* Arm B then Arm E

  * Arm B (induction): Patients receive rituximab IV on day 1; bortezomib IV on days 1, 4, 8, and 11; and bendamustine hydrochloride IV over 1 hour on days 1 and 4. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Arm E (continuation): Beginning 4 weeks after the completion of induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab as in arm D.
* Arm C then Arm F

  * Arm C (induction): Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Arm F (continuation): Immediately after completing induction therapy, patients who have stable disease or better at time of post-induction restaging receive oral lenalidomide on days 1-21. Treatment repeats every 4 weeks for 13 courses in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after the completion of induction therapy, these patients receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

Quality of life (including fatigue, neurotoxicity, anxiety, and depression) is assessed by questionnaire at baseline and periodically during study therapy.

Blood, bone marrow, and tissue samples may be collected periodically for correlative studies and for a repository.

After completion of study therapy, patients are followed up periodically for 15 years.

ELIGIBILITY:
Inclusion Criteria (Induction):

* Histologically confirmed (biopsy-proven) diagnosis of follicular B-cell non-Hodgkin lymphoma with no evidence of transformation to large cell histology

  * Patients having both diffuse and follicular architectural elements are eligible if the histology is predominantly follicular (i.e., ≥ 50% of the cross-sectional area) and there is no evidence of transformation to a large cell histology
  * Diagnostic confirmation (i.e., core needle or excisional lymph node biopsy) required if the interval since tissue diagnosis of low-grade malignant lymphoma is > 24 months

    * Bone marrow biopsy alone not acceptable
* Stage II, III, or IV AND grade 1, 2, or 3a disease
* Must meet criteria for High Tumor Burden (higher risk) as defined by either the Groupe D'Etude des Lymphomes Follicularies (GELF) criteria OR the follicular lymphoma international prognostic index (FLIPI) as defined below:

  * Patient must meet ≥ 1 of the following GELF criteria:

    * Nodal or extranodal mass ≥ 7 cm
    * At least 3 nodal masses > 3.0 cm in diameter
    * Systemic symptoms due to lymphoma or B symptoms
    * Splenomegaly with spleen > 16 cm by CT scan
    * Evidence of compression syndrome (e.g., ureteral, orbital, gastrointestinal) or pleural or peritoneal serous effusion due to lymphoma (irrespective of cell content)
    * Leukemic presentation (≥ 5.0 x 10^9/L malignant circulating follicular cells)
    * Cytopenias (polymorphonuclear leukocytes < 1.0 X 10^9/L, hemoglobin < 10 g/dL, and/or platelets < 100 x 10^9/L)
  * Patient must have a FLIPI-1 score of 3, 4, or 5 (1 point per criterion below):

    * Age ≥ 60 years
    * Stage III-IV disease
    * Hemoglobin level < 12 g/dL
    * > 4 nodal areas
    * Serum lactate dehydrogenase (LDH) level above normal
* At least 1 objective measurable disease parameter

  * Baseline measurements and evaluations (PET and CT) obtained within 6 weeks of randomization
  * Measurable disease in the liver is required if the liver is the only site of lymphoma
* HIV-positive patients must meet all of the following criteria:

  * HIV is sensitive to antiretroviral therapy
  * Must be willing to take effective antiretroviral therapy if indicated
  * No history of CD4 < 300 cells/mm³ prior to or at the time of lymphoma diagnosis
  * No history of AIDS-defining conditions
  * If on antiretroviral therapy, must not be taking zidovudine or stavudine
  * Must be willing to take prophylaxis for Pneumocystis jiroveci pneumonia (PCP) during therapy and ≥ 2 months following completion of study therapy or until the CD4 cells recover to over 250 cells/mm³
* ECOG performance status 0-2
* Absolute neutrophil count (ANC) ≥ 1,500/mm³ (includes neutrophils and bands)
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤ 5 x upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 x ULN
* Total bilirubin ≤ 1.5 x ULN (patients with known Gilbert disease should contact the study PI)
* Negative pregnancy test
* Fertile patients must use 2 effective methods (1 highly effective and 1 additional effective method) of contraception ≥ 28 days before, during, and for ≥ 28 days after completing study treatment
* Must register into the mandatory RevAssist® program and be willing and able to comply with the requirements of RevAssist® (for patients randomized to arm C and proceed onto arm F)

Exclusion Criteria (Induction):

* Prior chemotherapy, radiotherapy, or immunotherapy for lymphoma

  * Prednisone or other corticosteroids used for non-lymphomatous conditions will not be considered as prior chemotherapy
  * A prior/recent short course (< 2 weeks) of steroids for symptom relief of lymphoma-related symptoms is allowed
* Recent history of malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for ≥ 2 years
* Pregnant or nursing
* Active, uncontrolled infections (afebrile for > 48 hours off antibiotics)
* ≥ grade 2 neuropathy
* Myocardial infarction within the past 6 months
* NYHA class III-IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Known hypersensitivity to boron or mannitol
* Chronic carriers of hepatitis B virus (HBV) with positive hepatitis surface antigen (HBsAg +)

Inclusion Criteria (Continuation):

* Patient must have improved their response or have had no interval change in their tumor measurements with restaging from Induction cycle 3 to 6 as determined at Cycle 6 restaging.
* Adequate organ function
* ECOG performance status 0-2
* Patients with a prior history of HBV infection, but immune, with only IgG hepatitis core antibody positive (HBcAb+), must receive antiviral prophylaxis (e.g., lamivudine 100 mg po daily) for ≥ 1 week prior to course 1 and throughout induction and continuation therapy and for ≥ 12 months after the last rituximab dose
* Additional requirements for Arm C induction patients registering to arm F:

  * Patients must be willing to take deep vein thrombosis (DVT) prophylaxis. Subjects with a history of a thrombotic vascular event will be required to have full anticoagulation, therapeutic doses of low molecular weight heparin or warfarin to maintain an INR between 2.0 - 3.0, or any other accepted full anticoagulation regimen (e.g. direct thrombin inhibitors or Factor Xa inhibitors) with appropriate monitoring for that agent. Subjects without a history of a thromboembolic event are required to take a daily aspirin (81 mg or 325 mg) for DVT prophylaxis. Subjects who are unable to tolerate aspirin should receive low molecular weight heparin therapy or warfarin treatment or another accepted full anticoagulation regimen.
  * Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study/lenalidomide: 1) for at least 28 days before starting lenalidomide; 2) while participating in the study; and 3) for at least 28 days after discontinuation/stopping lenalidomide. The two methods of reliable contraception must include one highly effective method (i.e. intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and one additional effective (barrier) method (i.e. latex condom, diaphragm, cervical cap). FCBP must be referred to a qualified provider of contraceptive methods if needed.
  * Patient must agree to abstain from donating blood during study participation and for at least 28 days after discontinuation from protocol treatment.
  * All males, regardless of whether they have undergone a successful vasectomy, must agree to use a latex condom during sexual contact with a female of childbearing potential, or to practice complete abstinence from heterosexual intercourse with any female of childbearing potential during the cycles of continuation therapy of which lenalidomide are taken and for at least 28 days after discontinuation/stopping lenalidomide. Patient must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation from protocol treatment.
  * Must register into the mandatory RevAssist® program and be willing and able to comply with the requirements of RevAssist®

Exclusion Criteria (Continuation):

* Active, uncontrolled infections (afebrile for > 48 hours off antibiotics)
* ≥ grade 2 neuropathy
* Additional requirements for Arm C induction patients registering to arm F:

  * Not pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-02-09 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M. Evens, DO, MS, Principal Investigator — Robert H. Lurie Cancer Center
Locations (227):
- United States (227):
  - Marin Cancer Care Inc, Greenbrae, California
  - Salinas Valley Memorial, Salinas, California
  - Stanford University Hospitals and Clinics, Stanford, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Comprehensive Cancer Care and Research Institute of Colorado LLC, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Georgia Regents University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - IU Health Arnett Cancer Care, Lafayette, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Ottumwa Regional Health Center, Ottumwa, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Cancer Institute of New Jersey At Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - UMDNJ - New Jersey Medical School, Newark, New Jersey
  - New York University Langone Medical Center, New York, New York
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ireland Cancer Center Landerbrook Health Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - UHHS-Chagrin Highlands Medical Center, Orange, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - UH-Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology at Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Aria Health-Torresdale Campus, Philadelphia, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - West Virginia University Charleston, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology, Appleton, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Hematology and Oncology Clinic, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Oconomowoc Memorial Hospital-ProHealth Care Inc, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic, Two Rivers, Wisconsin
  - Waukesha Memorial Hospital - ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Evens AM, Hong F, Habermann TM, Advani RH, Gascoyne RD, Witzig TE, Quon A, Ranheim EA, Ansell SM, Cheema PS, Dy PA, O'Brien TE, Winter JN, Cescon TP, Chang JE, Kahl BS. A Three-Arm Randomized Phase II Study of Bendamustine/Rituximab with Bortezomib Induction or Lenalidomide Continuation in Untreated Follicular Lymphoma: ECOG-ACRIN E2408. Clin Cancer Res. 2020 Sep 1;26(17):4468-4477. doi: 10.1158/1078-0432.CCR-20-1345. Epub 2020 Jun 12. PMID 32532790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on December 13, 2010, accrued its first patient on February 9, 2011, and closed on May 13, 2015, with final accrual of 289 patients
Groups:
- Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab): Arm A (induction): Patients receive rituximab intravenously (IV) on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Arm D (continuation): Beginning 4 weeks after the completion of induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
  Bendamustin: Given IV
- Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab): Arm B (induction): Patients receive rituximab IV on day 1; bortezomib IV on days 1, 4, 8, and 11; and bendamustine hydrochloride IV over 1 hour on days 1 and 4. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Arm E (continuation): Beginning 4 weeks after the completion of induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab as in arm D.
  rituximab: Given IV
  Bendamustin: Given IV
  bortezomib: Given IV
- Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab): Arm C (induction): Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Arm F (continuation): Immediately after completing induction therapy, patients who have stable disease or better at time of post-induction restaging receive oral lenalidomide on days 1-21. Treatment repeats every 4 weeks for 13 courses in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after the completion of induction therapy, these patients receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  rituximab: Given IV
  Bendamustin: Given IV
  lenalidomide: Given orally
Period: Induction
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Started | 65 | 99 | 125
Received Treatment and Assessed for Toxicities | 65 | 93 | 122
Eligible and Treated | 59 | 85 | 114
Included in the Primary Analysis of Complete Remission Rate During Induction Treatment | 48 | 85 | 89
Completed | 61 | 80 | 104
Not Completed | 4 | 19 | 21
Not completed — Never started treatment | 0 | 6 | 3
Not completed — Lack of Efficacy | 4 | 3 | 7
Not completed — Adverse Event | 0 | 5 | 5
Not completed — Death | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 4 | 2
Not completed — Other disease | 0 | 1 | 2
Period: Continuation
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Started | 59 | 71 | 94
Received Continuation Treatment | 59 | 70 | 89
Completed | 44 | 56 | 51
Not Completed | 15 | 15 | 43
Not completed — Lack of Efficacy | 3 | 2 | 7
Not completed — Adverse Event | 5 | 3 | 16
Not completed — Death | 1 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 5 | 9
Not completed — Other diseases | 0 | 2 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Non-compliance | 1 | 0 | 1
Not completed — Insurance change | 0 | 1 | 0
Not completed — Mistakenly stayed on treatment for longer than expected | 0 | 1 | 0
Not completed — Not reported | 0 | 0 | 1
Not completed — Never started treatment | 0 | 1 | 5

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab) | Total
Number analyzed (Participants) | 59 | 85 | 114 | 258
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 79] | 60 [24 to 86] | 61 [24 to 88] | 61 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 34 | 56 | 116
  Male | 33 | 51 | 58 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 5 | 9
  Not Hispanic or Latino | 55 | 82 | 107 | 244
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 3 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 6 | 11
  White | 53 | 78 | 102 | 233
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate
Description: Complete remission is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy.
  This analysis was conducted among 222 evaluable patients for the primary analysis. The purpose of this analysis is to compare the complete remission rate of rituximab + bendamustine vs. bortezomib + rituximab + bendamustine as induction therapy, therefore, the proportion of patients with complete remission was compared between Arm B (bortezomib + rituximab + bendamustine) and Arms A and C combined (rituximab + bendamustine).
Time Frame: Assessed every 4 weeks during induction treatment and every 8 weeks during continuation treatment, up to 2 years
Population: This analysis was conducted among 222 evaluable patients for the primary analysis. The purpose of this analysis is to compare the complete remission rate of rituximab + bendamustine vs. bortezomib + rituximab + bendamustine as induction therapy, therefore, the proportion of patients with complete remission was compared between Arm B (bortezomib + rituximab + bendamustine) and Arms A and C combined (rituximab + bendamustine).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm A and Arm C (Induction With Bendamustine + Rituximab): Patients receive rituximab intravenously (IV) on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm B (Induction With Bendamustine + Rituximab + Bortezomib): Patients receive rituximab IV on day 1; bortezomib IV on days 1, 4, 8, and 11; and bendamustine hydrochloride IV over 1 hour on days 1 and 4. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A and Arm C (Induction With Bendamustine + Rituximab) | Arm B (Induction With Bendamustine + Rituximab + Bortezomib)
Number analyzed (Participants) | 137 | 85
proportion of participants | 0.62 [0.53 to 0.70] | 0.75 [0.65 to 0.84]
Statistical Analysis 1: Comparison: Arm A and Arm C (Induction With Bendamustine + Rituximab) vs Arm B (Induction With Bendamustine + Rituximab + Bortezomib); The study was designed to detect a 16% difference in CR rate from 50% in the Bendamustine + Rituximab arms to 66% in the Bendamustine + Rituximab + Bortezomib arm, with 90% power at the one-sided alpha 0.15 level; Test type: Superiority; p = 0.02, Cochran-Mantel-Haenszel — one-sided p-value

2. Primary Outcome: 1-year Post-induction Disease-free Survival (DFS) Rate
Description: 1-year post induction disease-free survival rate is defined as the proportion of patients achieving complete remission during induction treatment and are alive and maintaining complete remission at 1 year after induction completion.
  The purpose of this analysis is to compare the 1-year post-induction disease-free survival (DFS) rate with rituximab plus lenalidomide to rituximab alone as continuation therapy following induction treatment of bendamustine+rituximab, therefore, patients with induction treatment of bendamustine + rituximab + bortezomib were not included in this analysis.
Time Frame: Assessed at 1 year post-induction, approximately 1.5 years
Population: All eligible and treated patients in the continuation phase of arm A + D and arm C + F.
  The purpose of this analysis is to compare the 1-year post-induction disease-free survival (DFS) rate with rituximab plus lenalidomide to rituximab alone as continuation therapy following induction treatment of bendamustine+rituximab, therefore, patients with induction treatment of bendamustine + rituximab + bortezomib were not included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 53 | 84
proportion of participants | 0.85 [0.72 to 0.93] | 0.67 [0.56 to 0.77]
Statistical Analysis 1: Comparison: Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) vs Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab); Test type: Superiority; p = 0.02, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified on Groupe d'Etude des Lymphomes Folliculaires status and Follicular Lymphoma International Prognostic Index

3. Secondary Outcome: 3-year Progression-free Survival Rate
Description: Progression-free survival is defined as the time from registration of induction treatment to progression, relapse or death, whichever occurs first. Patients alive without documented progression are censored at last disease assessment. 3-year progression-free survival rate is the proportion of patients who were progression-free and alive at 3 years estimated using the method of Kaplan-Meier.
  Progression/relapse is defined as appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, >=50% increase from nadir in the SPD of any previously involved nodes or extranodal masses or the size of other lesions, or >=50% increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in its short axis.
Time Frame: Assessed every cycle during treatment and every 6 months between 2 and 5 years from study entry
Population: This analysis was conducted among 222 evaluable patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 48 | 85 | 89
proportion of participants | 0.77 [0.65 to 0.90] | 0.82 [0.74 to 0.91] | 0.76 [0.67 to 0.85]

4. Secondary Outcome: 5-year Overall Survival Rate
Description: Overall survival is defined as the time from randomization to death or date last known alive. 5-year overall survival rate is the proportion of patients who were alive at 5 years estimated using the method of Kaplan-Meier.
Time Frame: Assessed every cycle during treatment and every 6 months between 2 and 5 years from study entry
Population: This analysis was conducted among 222 evaluable patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 48 | 85 | 89
proportion of participants | 0.87 [0.79 to 0.97] | 0.86 [0.77 to 0.94] | 0.83 [0.75 to 0.91]

5. Secondary Outcome: Complete Remission (CR) Rate
Description: Complete remission is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy.
  This analysis was conducted among 222 evaluable patients. The proportion of patients with complete remission was compared between patients with Follicular Lymphoma International Prognostic Index (FLIPI) of 3-5 and patients with FLIPI of 0-2/unknown.
  The FLIPI was developed in order to predict prognosis of patients with newly diagnosed follicular lymphoma (FL). The five FLIPI risk factors were: age > 60 years, Ann Arbor stage III-IV, hemoglobin level < 12 gm/dL, >4 nodal areas, and serum LDH level above normal. The FLIPI score was calculated by summing the number of risk factors. The higher the FLIPI score, the worse the prognosis.
Time Frame: Assessed every 4 weeks during induction treatment and every 8 weeks during continuation treatment, up to 2 years
Population: This analysis was conducted among 222 evaluable patients that were enrolled before activation of addendum #8. The proportion of patients with complete remission was compared between FLIPI 0-2/unknown and FLIPI 3-5 at baseline.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- FLIPI 0-2/Unknown: Patients with baseline follicular lymphoma international prognostic index (FLIPI) score of 0-2 or unknown.
- FLIPI 3-5: Patients with baseline follicular lymphoma international prognostic index (FLIPI) score of 3-5.
Arm/Group | FLIPI 0-2/Unknown | FLIPI 3-5
Number analyzed (Participants) | 101 | 121
proportion of participants | 0.71 [0.61 to 0.80] | 0.64 [0.54 to 0.72]

6. Secondary Outcome: 1-year Disease-free Survival (DFS) Rate
Description: 1-year post induction disease-free survival rate is defined as the proportion of patients achieving complete remission during induction treatment and are alive and maintaining complete remission at 1 year after induction completion.
  This analysis was conducted among 203 evaluable patients in the continuation treatment portion of the study. The 1-year post induction disease-free survival rate was compared between patients with FLIPI of 3-5 and patients with FLIPI of 0-2/unknown.
  The FLIPI was developed in order to predict prognosis of patients with newly diagnosed follicular lymphoma (FL). The five FLIPI risk factors were: age > 60 years, Ann Arbor stage III-IV, hemoglobin level < 12 gm/dL, >4 nodal areas, and serum LDH level above normal. The FLIPI score was calculated by summing the number of risk factors. The higher the FLIPI score, the worse the prognosis.
Time Frame: Assessed at 1 year post-induction, approximately 1.5 years
Population: This analysis was conducted among 203 evaluable patients in the continuation treatment portion of the study. The 1-year post induction disease-free survival rate was compared between patients with FLIPI of 3-5 and patients with FLIPI of 0-2/unknown.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLIPI 0-2/Unknown | FLIPI 3-5
Number analyzed (Participants) | 91 | 112
proportion of participants | 0.84 [0.74 to 0.90] | 0.74 [0.65 to 0.82]

7. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is defined as the time from registration of induction treatment to progression, relapse or death, whichever occurs first. Patients alive without documented progression are censored at last disease assessment. Progression/relapse is defined as appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, >=50% increase from nadir in the SPD of any previously involved nodes or extranodal masses or the size of other lesions, or >=50% increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in its short axis.
  The five FLIPI risk factors were: age > 60 years, Ann Arbor stage III-IV, hemoglobin level < 12 gm/dL, >4 nodal areas, and serum LDH level above normal. The FLIPI score was calculated by summing the number of risk factors. The higher the FLIPI score, the worse the prognosis.
Time Frame: Assessed every cycle during treatment and every 6 months between 2 and 5 years from study entry
Population: This analysis was conducted among 222 evaluable patients that were enrolled before activation of addendum #8.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | FLIPI 0-2/Unknown | FLIPI 3-5
Number analyzed (Participants) | 101 | 121
years | 6.1 [6.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 6.2 [4.5 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

8. Secondary Outcome: 5-year Overall Survival Rate
Description: Overall survival is defined as the time from randomization to death or date last known alive. 5-year overall survival rate is the proportion of patients who were alive at 5 years estimated using the method of Kaplan-Meier.
  The FLIPI was developed in order to predict prognosis of patients with newly diagnosed follicular lymphoma (FL). The five FLIPI risk factors were: age > 60 years, Ann Arbor stage III-IV, hemoglobin level < 12 gm/dL, >4 nodal areas, and serum LDH level above normal. The FLIPI score was calculated by summing the number of risk factors. The higher the FLIPI score, the worse the prognosis.
Time Frame: Assessed every cycle during treatment and every 6 months between 2 and 5 years from study entry
Population: This analysis was conducted among 222 evaluable patients.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | FLIPI 0-2/Unknown | FLIPI 3-5
Number analyzed (Participants) | 101 | 121
proportion of participants | 0.90 [0.84 to 0.96] | 0.81 [0.74 to 0.89]

9. Secondary Outcome: Complete Remission (CR) Rate
Description: Complete remission is defined as complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present prior to therapy.
  This analysis was conducted among 250 evaluable patients with Cumulative Illness Rating Scale (CIRS) data available. The proportion of patients with complete remission was compared between patients with CIRS <10 and patients with CIRS >=10. Higher CIRS scores indicate higher severity with max score of 56 points.
Time Frame: Assessed every 4 weeks during induction treatment and every 8 weeks during continuation treatment, up to 2 years
Population: This analysis was conducted among 250 evaluable patients with baseline CIRS data available. The proportion of patients with complete remission was compared between baseline CIRS <10 and baseline CIRS >=10.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- CIRS <10: Patients with baseline Cumulative Illness Rating Scale (CIRS) score <10
- CIRS >=10: Patients with baseline Cumulative Illness Rating Scale (CIRS) score >=10
Arm/Group | CIRS <10 | CIRS >=10
Number analyzed (Participants) | 207 | 43
proportion of participants | 0.70 [0.63 to 0.76] | 0.70 [0.54 to 0.83]

10. Secondary Outcome: 1-year Disease-free Survival (DFS) Rate
Description: 1-year post induction disease-free survival rate is defined as the proportion of patients achieving complete remission during induction treatment and are alive and maintaining complete remission at 1 year after induction completion.
  This analysis was conducted among 250 evaluable patients with Cumulative Illness Rating Scale (CIRS) data available. The proportion of patients disease-free and alive at 1 year post induction treatment was compared between patients with CIRS <10 and patients with CIRS >=10. Higher CIRS scores indicate higher severity with max score of 56 points.
Time Frame: Assessed at 1 year post-induction, approximately 1.5 years
Population: This analysis was conducted among 250 evaluable patients with baseline Cumulative Illness Rating Scale (CIRS) data available. The proportion of patients disease-free and alive at 1 year post induction treatment was compared between patients with CIRS <10 and patients with CIRS >=10.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CIRS <10 | CIRS >=10
Number analyzed (Participants) | 207 | 43
proportion of participants | 0.62 [0.55 to 0.69] | 0.65 [0.49 to 0.79]

11. Secondary Outcome: 3-year Progression-free Survival Rate
Description: Progression-free survival is defined as the time from registration of induction treatment to progression, relapse or death, whichever occurs first. Patients alive without documented progression are censored at last disease assessment. 3-year progression-free survival rate is the proportion of patients who were progression-free and alive at 3 years estimated using the method of Kaplan-Meier.
  Progression/relapse is defined as appearance of any new lesion more than 1.5 cm in any axis during or at the end of therapy, >=50% increase from nadir in the SPD of any previously involved nodes or extranodal masses or the size of other lesions, or >=50% increase in the longest diameter of any single previously identified node or extranodal mass more than 1 cm in its short axis.
  The 3-year progression-free survival rate is reported by Cumulative Illness Rating Scale (CIRS) score (<10 vs. >=10). Higher CIRS scores indicate higher severity with max score of 56 points.
Time Frame: Assessed every cycle during treatment and every 6 months between 2 and 5 years from study entry
Population: This analysis was conducted among 250 evaluable patients with baseline Cumulative Illness Rating Scale (CIRS) data available.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CIRS <10 | CIRS >=10
Number analyzed (Participants) | 207 | 43
proportion of participants | 0.83 [0.77 to 0.88] | 0.68 [0.54 to 0.85]

12. Secondary Outcome: 5-year Overall Survival Rate
Description: Overall survival is defined as the time from randomization to death or date last known alive. 5-year overall survival rate is the proportion of patients who were alive at 5 years estimated using the method of Kaplan-Meier.
  The 5-year overall survival rate is reported by Cumulative Illness Rating Scale (CIRS) score (<10 vs. >=10). Higher CIRS scores indicate higher severity with max score of 56 points.
Time Frame: Assessed every cycle during treatment and every 6 months between 2 and 5 years from study entry
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | CIRS <10 | CIRS >=10
Number analyzed (Participants) | 207 | 43
proportion of participants | 0.87 [0.83 to 0.92] | 0.80 [0.69 to 0.94]

13. Secondary Outcome: Proportion of Patients With Grade 3 or Higher Peripheral Neuropathy
Description: Peripheral neuropathy was assessed using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Proportion of patients with grade 3 or higher peripheral neuropathy was compared between patients with subcutaneous bortezomib and patients with intravenous bortezomib.
Time Frame: Assessed every cycle during treatment and for 30 days after discontinuation of treatment, up to 15 years
Population: This analysis was conducted among 99 patients who received bortezomib.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Subcutaneous Bortezomib: Patients who received subcutaneous bortezomib.
- Intravenous Bortezomib: Patients who received intravenous bortezomib. Patients who received both subcutaneous and intravenous bortezomib are included in the intravenous bortezomib group.
Arm/Group | Subcutaneous Bortezomib | Intravenous Bortezomib
Number analyzed (Participants) | 17 | 82
proportion of participants | 0.06 [0.002 to 0.29] | 0.12 [0.06 to 0.21]

14. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G) Total Score at Baseline
Description: The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire that has four areas of measurements (physical well-being, social/family well-being, emotional well-being and functional well-being) with a scale of 0-4. The FACT-G total score ranges between 0 and 108. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline
Population: All enrolled patients with baseline FACT-G total score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 63 | 91 | 119
score on a scale | 83.9 (14.2) | 84.7 (15.5) | 86.0 (16.0)

15. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G) Total Score at Mid-treatment
Description: The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire that has four areas of measurements (physical well-being, social/family well-being, emotional well-being and functional well-being) with a scale of 0-4. The FACT-G total score ranges between 0 and 108. The higher the score, the better the quality of life.
  FACT-G total score at cycle 3 is considered as mid-treatment score. If FACT-G total score at cycle 3 is not available, the score at cycle 4 will be used as the mid-treatment score.
Time Frame: Assessed at cycle 3 or cycle 4, approximately 3 or 4 months
Population: All enrolled patients with cycle 3 or cycle 4 FACT-G total score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 55 | 74 | 107
score on a scale | 85.5 (15.7) | 84.2 (16.4) | 85.2 (15.9)

16. Secondary Outcome: Functional Assessment of Cancer Therapy - General (FACT-G) Total Score at End of Induction Treatment
Description: as for outcome 14
Time Frame: Assessed at cycle 6, approximately 6 months
Population: All enrolled patients with cycle 6 FACT-G total score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 54 | 71 | 101
score on a scale | 86.0 (17.7) | 86.5 (13.9) | 84.9 (18.2)

17. Secondary Outcome: Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Subscale Score at Baseline
Description: The Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) is a 15-item questionnaire that evaluates disease-related symptoms and concerns specific to lymphoma with a scale of 0-4. The FACT-Lym subscale score ranges between 0 and 60. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline
Population: All enrolled patients with baseline FACT-Lym subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 63 | 91 | 120
score on a scale | 43.8 (8.7) | 44.3 (9.3) | 44.9 (10.6)

18. Secondary Outcome: Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Subscale Score at Mid-induction Treatment
Description: The Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) is a 15-item questionnaire that evaluates disease-related symptoms and concerns specific to lymphoma with a scale of 0-4. The FACT-Lym subscale score ranges between 0 and 60. The higher the score, the better the quality of life.
  FACT-Lym subscale score at cycle 3 is considered as mid-treatment score. If FACT-Lym subscale score at cycle 3 is not available, the score at cycle 4 will be used as the mid-treatment score.
Time Frame: Assessed at cycle 3 or cycle 4, approximately 3 or 4 months
Population: All enrolled patients with cycle 3 or cycle 4 FACT-Lym subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 55 | 75 | 108
score on a scale | 47.9 (7.4) | 46.8 (8.7) | 46.5 (9.5)

19. Secondary Outcome: Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) Subscale Score at End of Induction Treatment
Description: as for outcome 17
Time Frame: Assessed at cycle 6, approximately 6 months
Population: All enrolled patients with cycle 6 FACT-Lym subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 54 | 71 | 101
score on a scale | 48.9 (7.5) | 48.4 (8.5) | 47.2 (9.9)

20. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Subscale Score at Baseline
Description: The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) is comprised of 13 items that assess fatigue and its impact with a scale of 0-4. The FACIT-Fatigue subscale score ranges between 0 and 52. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline
Population: All enrolled patients with baseline FACIT-Fatigue subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 63 | 91 | 120
score on a scale | 38.6 (10.5) | 37.9 (11.4) | 38.1 (12.1)

21. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Subscale Score at Mid-induction Treatment
Description: The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) is comprised of 13 items that assess fatigue and its impact with a scale of 0-4. The FACIT-Fatigue subscale score ranges between 0 and 52. The higher the score, the better the quality of life.
  FACIT-Fatigue subscale score at cycle 3 is considered as mid-treatment score. If FACIT-Fatigue subscale score at cycle 3 is not available, the score at cycle 4 will be used as the mid-treatment score.
Time Frame: Assessed at cycle 3 or cycle 4, approximately 3 or 4 months
Population: All enrolled patients with cycle 3 or cycle 4 FACIT-Fatigue subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 55 | 75 | 108
score on a scale | 39.2 (9.0) | 34.5 (10.9) | 36.3 (12.3)

22. Secondary Outcome: Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-Fatigue) Subscale Score at End of Induction Treatment
Description: as for outcome 20
Time Frame: Assessed at cycle 6, approximately 6 months
Population: All enrolled patients with cycle 6 FACIT-Fatigue subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 54 | 71 | 100
score on a scale | 39.9 (10.1) | 39.1 (9.8) | 36.3 (12.2)

23. Secondary Outcome: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT-GOG-NTX) Subscale Score at Baseline
Description: The Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT-GOG-NTX) subscale is comprised of 11 items that assess neurotoxicity with a scale of 0-4. The FACT-GOG-NTX subscale score ranges between 0 and 44. The higher the score, the better the quality of life.
Time Frame: Assessed at baseline
Population: All enrolled patients with baseline FACT-GOG-NTX subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 46 | 65 | 90
score on a scale | 39.9 (4.3) | 38.7 (6.0) | 38.8 (5.5)

24. Secondary Outcome: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT-GOG-NTX) Subscale Score at Mid-induction Treatment
Description: as for outcome 23
Time Frame: Assessed at cycle 3, approximately 3 months
Population: All enrolled patients with cycle 3 FACT-GOG-NTX subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 58 | 80 | 109
score on a scale | 40.0 (4.6) | 38.6 (5.1) | 39.1 (5.2)

25. Secondary Outcome: Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT-GOG-NTX) Subscale Score at the End of Induction Treatment
Description: as for outcome 23
Time Frame: Assessed at end of induction treatment (cycle 6), approximately 6 months
Population: All enrolled patients with cycle 6 FACT-GOG-NTX subscale score available
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A Then Arm D (Induction With Bendamustine + Rituximab; Continuation With Rituximab) | Arm B Then Arm E (Induction With Bendamustine + Rituximab + Bortezomib; Continuation With Rituximab) | Arm C Then Arm F (Induction With Bendamustine+Rituximab; Continuation With Lenalidomide + Rituximab)
Number analyzed (Participants) | 52 | 69 | 96
score on a scale | 39.8 (4.0) | 36.1 (6.5) | 39.0 (5.9)

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment, up to 5 years
Description: Serious Adverse Events include post-baseline adverse events of grade 3 and higher that are definitely, probably or possibly related to protocol treatment based on the case report forms (CRFs).
  Only patients who started protocol therapy are included in the analysis of adverse events. All registered patients are included in the analysis of all-cause mortality.
  Deaths were counted in Step 1 (Arms A, B and C) for patients who did not registered to Step 2 continuation treatment.
Groups:
- Arm A: Arm A (induction): Patients receive rituximab intravenously (IV) on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm B: Arm B (induction): Patients receive rituximab IV on day 1; bortezomib IV on days 1, 4, 8, and 11; and bendamustine hydrochloride IV over 1 hour on days 1 and 4. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm C: Arm C (induction): Patients receive rituximab IV on day 1 and bendamustine hydrochloride IV over 1 hour on days 1 and 2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
- Arm D: Arm D (continuation after Arm A): Beginning 4 weeks after the completion of Arm A induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
- Arm E: Arm E (continuation after Arm B): Beginning 4 weeks after the completion of Arm B induction therapy, patients who have stable disease or better at time of post-induction restaging receive rituximab as in arm D.
- Arm F: Arm F (continuation after Arm C): Immediately after completing Arm C induction therapy, patients who have stable disease or better at time of post-induction restaging receive oral lenalidomide on days 1-21. Treatment repeats every 4 weeks for 13 courses in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after the completion of induction therapy, these patients receive rituximab IV on day 1. Treatment repeats every 8 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E | Arm F
All-Cause Mortality (participants affected / at risk) | 2/65 | 9/99 | 12/125 | 6/59 | 7/71 | 10/94
Serious Adverse Events (participants affected / at risk) | 51/65 | 78/93 | 96/122 | 39/59 | 44/70 | 77/89
Other Adverse Events (participants affected / at risk) | 64/65 | 92/93 | 122/122 | 59/59 | 70/70 | 88/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=65) | Arm B (N=93) | Arm C (N=122) | Arm D (N=59) | Arm E (N=70) | Arm F (N=89)
Anemia (Blood and lymphatic system disorders) | 2 | 3 | 5 | 0 | 1 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 6 | 1 | 2 | 9
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Blood and lymphatic disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 6 | 9 | 1 | 0 | 5
Fever (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 1 | 3 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 3 | 0 | 1 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 6 | 2 | 1 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 4 | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 1 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 2 | 1 | 0 | 0 | 1
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bladder infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 3 | 0 | 1 | 0 | 7
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral nerve infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Skin infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Cholesterol high (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 44 | 61 | 77 | 33 | 35 | 56
Neutrophil count decreased (Investigations) | 22 | 33 | 35 | 12 | 13 | 58
Platelet count decreased (Investigations) | 2 | 9 | 7 | 0 | 2 | 2
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 1 | 2 | 0 | 1 | 0
White blood cell decreased (Investigations) | 19 | 32 | 30 | 14 | 11 | 52
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 3 | 0 | 0 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 11 | 1 | 0 | 3 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 3 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 2 | 3 | 2 | 1 | 2
Hypotension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 2
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=65) | Arm B (N=93) | Arm C (N=122) | Arm D (N=59) | Arm E (N=70) | Arm F (N=89)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 3 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 39 | 59 | 67 | 32 | 35 | 54
Chills (General disorders) | 3 | 16 | 8 | 1 | 1 | 10
Edema limbs (General disorders) | 5 | 14 | 16 | 6 | 7 | 15
Fatigue (General disorders) | 53 | 74 | 92 | 38 | 51 | 67
Fever (General disorders) | 9 | 20 | 10 | 3 | 2 | 5
Infusion related reaction (General disorders) | 12 | 7 | 13 | 0 | 0 | 0
Injection site reaction (General disorders) | 3 | 8 | 3 | 0 | 0 | 0
Pain (General disorders) | 2 | 5 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 10 | 15 | 2 | 3 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 8 | 12 | 4 | 2 | 13
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 21 | 24 | 8 | 2 | 22
Abdominal pain (Gastrointestinal disorders) | 5 | 12 | 7 | 2 | 4 | 8
Constipation (Gastrointestinal disorders) | 22 | 45 | 46 | 7 | 7 | 27
Diarrhea (Gastrointestinal disorders) | 20 | 44 | 27 | 10 | 11 | 34
Dry mouth (Gastrointestinal disorders) | 2 | 7 | 9 | 0 | 3 | 9
Dyspepsia (Gastrointestinal disorders) | 7 | 8 | 13 | 5 | 2 | 6
Mucositis oral (Gastrointestinal disorders) | 6 | 7 | 19 | 1 | 0 | 6
Nausea (Gastrointestinal disorders) | 37 | 56 | 74 | 10 | 8 | 26
Vomiting (Gastrointestinal disorders) | 11 | 25 | 28 | 2 | 3 | 10
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 7 | 3 | 0 | 1 | 5
Allergic reaction (Immune system disorders) | 4 | 6 | 8 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 2 | 5 | 4
Peripheral nerve infection (Infections and infestations) | 0 | 0 | 0 | 3 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 3 | 6 | 5
Upper respiratory infection (Infections and infestations) | 3 | 3 | 7 | 2 | 3 | 14
Alanine aminotransferase increased (Investigations) | 12 | 19 | 13 | 8 | 13 | 14
Alkaline phosphatase increased (Investigations) | 9 | 12 | 10 | 3 | 6 | 11
Aspartate aminotransferase increased (Investigations) | 12 | 20 | 16 | 8 | 17 | 14
Blood bilirubin increased (Investigations) | 4 | 3 | 3 | 4 | 3 | 5
Creatinine increased (Investigations) | 5 | 6 | 7 | 5 | 4 | 11
Lymphocyte count decreased (Investigations) | 35 | 55 | 62 | 39 | 54 | 65
Neutrophil count decreased (Investigations) | 26 | 46 | 47 | 25 | 30 | 61
Platelet count decreased (Investigations) | 26 | 65 | 65 | 18 | 21 | 48
Weight loss (Investigations) | 10 | 20 | 24 | 5 | 8 | 5
White blood cell decreased (Investigations) | 42 | 60 | 78 | 39 | 45 | 78
Investigations - Other, specify (Investigations) | 4 | 4 | 5 | 3 | 11 | 5
Anorexia (Metabolism and nutrition disorders) | 17 | 34 | 46 | 8 | 6 | 21
Dehydration (Metabolism and nutrition disorders) | 3 | 8 | 7 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 14 | 10 | 9 | 14 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 16 | 13 | 2 | 2 | 12
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 14 | 12 | 2 | 4 | 10
Hypokalemia (Metabolism and nutrition disorders) | 6 | 12 | 12 | 4 | 1 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 4 | 5 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 5 | 13 | 8 | 0 | 5 | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 13 | 8 | 4 | 8 | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 8 | 10 | 2 | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 12 | 7 | 5 | 7 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 18 | 7 | 2 | 9 | 4
Musculoskeletal and connective - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 5
Dizziness (Nervous system disorders) | 6 | 13 | 12 | 2 | 1 | 9
Dysgeusia (Nervous system disorders) | 8 | 14 | 20 | 1 | 5 | 11
Headache (Nervous system disorders) | 9 | 21 | 15 | 3 | 3 | 11
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 4 | 2 | 4
Peripheral motor neuropathy (Nervous system disorders) | 2 | 8 | 3 | 3 | 7 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 15 | 61 | 24 | 15 | 42 | 22
Blurred vision (Eye disorders) | 0 | 6 | 2 | 1 | 4 | 3
Insomnia (Psychiatric disorders) | 5 | 11 | 14 | 4 | 3 | 8
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 11 | 3 | 8 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 15 | 16 | 5 | 5 | 14
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 4 | 4
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 1
Hypertension (Vascular disorders) | 1 | 7 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 10 | 4 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 4 | 1 | 4 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT01216683/Prot_SAP_000.pdf